CLINICAL TRIAL: NCT05231512
Title: The Effects of a Music Therapy Respiratory Protocol on Post-Covid Respiratory Symptoms
Brief Title: The Effects of a Music Therapy Respiratory Protocol on Post-Covid-19 Respiratory Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Joanne Loewy, Associate Clinical Professor, Director Louis Armstrong Dept. of Music & Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY 20-02110
Record Dates: First submitted 2022-02-07; First posted 2022-02-09 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Post Covid-19 Respiratory; Dyspnea; SARS-CoV 2
Keywords: Post-Covid-19; respiratory; pulmonary; music; therapy; music therapy
MeSH Terms: conditions — Dyspnea | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Individuals living with post-Covid-19 respiratory symptoms (Experimental): Live virtual music therapy interventions for people experiencing difficulties breathing after having had COVID-19 (diagnosed or presumed).
  Interventions: Other: Respiratory Music Therapy Protocol

INTERVENTIONS:
Other: Respiratory Music Therapy Protocol — Participants will engage in eight (8) 45-minute virtual music therapy groups containing up to 6 participants over the course of 8 weeks. Within these groups, participants will be invited to use instruments provided including a Yamaha recorder and a Grover Trophy slide whistle. 45 minute virtual music therapy sessions facilitated by board-certified music therapy will consist of music-assisted relaxation through music visualization, followed by gentle pulmonary exercise via wind instrumental playing, and concluding with group singing.
  Other Names: Music therapy

SUMMARY:
The effects of a tested and published music therapy respiratory protocol shown to be efficacious with pediatric asthma and adult COPD is being studied with individuals living with post-Covid-19 respiratory symptoms. An interventional, single arm study is being conducted with individuals meeting eligibility criteria detailed below. Primary outcome is a change in the MRC Dyspnea score, with secondary aims focusing on improved quality of life, including reduced fatigue and depression and improved sleep and resilience.

DETAILED DESCRIPTION:
Since November 2019, the SARS-CoV-2 (COVID-19) virus has rapidly spread to countries across the globe. The COVID-19 pandemic is particularly destructive in the U.S., where, as of August 2020, total case numbers exceed 4 million. Recovering patients of COVID-19 report symptoms of fatigue, dyspnea (shortness of breath) and other pulmonary dysfunctions. A study conducted in Italy, where cases spiked to around 40,000 in March, showed that 87.4% of participants with post-acute COVID-19 experience at least one persistent symptom. Pulmonologists facing the pressing challenge of creating a respiratory rehabilitation program for recovering COVID-19 patients can benefit from integrating music therapy into their practice. Music therapy is the use of music, vocal or instrumental, to therapeutically address the holistic needs of a patient. Several studies have been conducted in the past investigating the neurological and physiological benefits of music therapy for patients engaging in breath regulation, and with pulmonary dysfunction such as COPD or asthma. At Mount Sinai Beth Israel, the Louis Armstrong Department of Music Therapy provides the Music for AIR (Advances in Respiration) programs to treat patients with lung disease, especially those with COPD. Music for AIR has successfully used wind instrument playing, singing, and music visualization to ease common symptoms of COPD including dyspnea and fatigue. As dyspnea and fatigue are also common persisting symptoms of patients recovering from COVID-19, Music for AIR interventions and its possible therapeutic benefits for recovering COVID-19 patients warrant a necessary investigation. Currently, there is no research looking specifically at music therapy as a modality of treatment for physical symptoms in post-COVID-19 patients. Thus, the aim of this study is to utilized previously validated interventions to measure efficacy in this unique population.COVID-19 affects multiple organs and systems. Current evidence shows that effects of the virus have surpassed the acute phase, manifesting in residual symptoms in neurological, physical, cognitive, pulmonary, and emotional areas. Music therapy is a clinical therapy that has demonstrated efficacy in improving function in these aforementioned areas. The purpose of this study is to examine clinical music therapy - specifically including wind playing, singing, and music visualizations - to study the effects on physical function and quality of life for adults experiencing shortness of breath who have been previously diagnosed with (or presumptive) COVID-19. This study aims to test a previously studied music therapy protocol on patients presenting with continued respiratory symptoms following confirmed or presumed COVID-19 diagnosis over an 8-week period within a virtual group setting. Secondary aims to be monitored are any changes in depression, anxiety, fatigue, sleep, quality of life, and resilience.

ELIGIBILITY:
Inclusion Criteria:

* Participation in Mount Sinai Post-COVID Treatment Center care
* Confirmed or presumptive COVID-19 history based on symptoms
* Experiencing residual pulmonary issues (shortness of breath, fatigue)
* MRC Dyspnea score of grade 3, 4, or 5
* 18 years or older

Exclusion Criteria:

* Under 18 years
* MRC Dyspnea Score of grade 1 or 2
* Presence of respiratory issues without confirmed or presumptive COVID-19 diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
MRC dyspnea score | 12 weeks
  MRC Dyspnea Score -Total scale from 1-5, with higher score indicating more perceived breathlessness.

SECONDARY OUTCOMES:
Self-reported Chronic Respiratory Questionnaire (CRQ-SR) | 12 weeks
  20 item questionnaire, each item score from 1 to 7. Total range from 20-140, with higher score indicating better health outcomes.
Visual Analog Scale (VAS) | 12 weeks
  VAS full range from 0-10, with higher score indicating more fatigue
Beck Depression Inventory - short form (BDI-SF) | 12 weeks
  13 items, full range from 0-39, with higher score indicating more severe symptoms of depression.
General Anxiety Disorder 7-item questionnaire (GAD-7) | 12 weeks
  The General Anxiety Disorder 7-item questionnaire (GAD-7) is a 7-item questionnaire that asks user to rank how often they have been bothered by seven problems over the past two weeks from "0" (not at all) to "3" (nearly every day). Full scale from 0-21, with higher score indicating more symptoms.
Hospital Anxiety and Depression Scale (HADS) | 12 weeks
  Questionnaire with 7 items for anxiety and 7 items for depression, each item is scored on a 4 point response 0 - 3, scores for each subscale from 0 (normal) to 21 (severe symptoms) with full range from 0 to 42. Higher score indicating more distress.
Coronavirus Anxiety Scale (CAS) | 12 weeks
  5-item scale, each item scored 0 (not at all) to 4 (nearly every day over the last 2 weeks). Full scale from 0-20, with higher score indicating poorer health outcomes.
Fatigue Severity Scale | 12 weeks
  9 item scale, each item scored from 1 (strongly disagree) to 7 (strongly agree). Total scale from 9-63, with higher score indicating greater fatigue.
The Epworth Sleepiness Scale (ESS | 12 weeks
  An 8-item measure that asks about the probability of dozing or sleeping during typical daytime activities. Each item is scored from 0, no chance of dozing, to 3, high chance of dozing. Total scale from 0 to 24, with higher score indicating severe excessive daytime sleepiness.
EuroQoL 5 dimensions 5 levels (EQ-5D-5L) | 12 weeks
  The EQ-5D is a generic instrument for describing and valuing health. The new version includes the 5 levels of severity in each of the existing five EQ-5D dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, and now called the EQ-5D-5L. Full scale from 5 to 25, with higher score indicating poorer health outcomes.
Connor-davidson Resilience Scale (CD-RISC) | 12 weeks
  Self-report 25-item scale, each item score from 0 (not true at all) to 4 (true nearly all the time). Full scale from 0-100, with higher score indicating better health outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne V Loewy, DA, Principal Investigator — Director Louis Armstrong Center for Music & Medicine,
Locations (2):
- United States (2):
  - Louis Armstrong Dept. of Music & Medicine, Mount Sinai Union Square, New York, New York
  - NYC Health & Hospitals - Elmhurst, New York, New York

IPD SHARING:
Plan to Share IPD: No
The data is specific to this study only

REFERENCES:
- [Background] Loewy J, Goldsmith C, Deshpande S, Sun A, Harris J, van Es C, Zvi ZB, Dahmer S. Music therapy in pediatric asthma improves pulmonary function while reducing hospitalizations. J Asthma. 2021 May;58(5):674-682. doi: 10.1080/02770903.2020.1712725. Epub 2020 Jan 23. PMID 31906748
- [Background] Canga B, Azoulay R, Raskin J, Loewy J. AIR: Advances in Respiration - Music therapy in the treatment of chronic pulmonary disease. Respir Med. 2015 Dec;109(12):1532-9. doi: 10.1016/j.rmed.2015.10.001. Epub 2015 Oct 19. PMID 26522499